CLINICAL TRIAL: NCT05011318
Title: Effects of Cognitive Fatigue on Heart Rate Variability and Skin Conductance
Acronym: FRESH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanyang Technological University (Other)
Collaborators: National Research Foundation, Singapore (Other Government); Ministry of National Development, Singapore (Other Government); Housing and Development Board, Singapore (Other Government)
Responsible Party: Principal Investigator, Georgios CHRISTOPOULOS, Associate Professor, Nanyang Technological University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COT-V4-2020-1-S002
Record Dates: First submitted 2021-08-12; First posted 2021-08-18 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Cognitive Fatigue; Mental Fatigue; Behavioral Performance; Heart Rate Variability; Skin Conductance
MeSH Terms: conditions — Mental Fatigue | interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fatigue Manipulation (Experimental)
  Interventions: Other: Baseline; Other: Fatigue Manipulation

INTERVENTIONS:
Other: Baseline — 5-min urban park video clip (Presented on a TV)
Other: Fatigue Manipulation — 20-min 2-back task (Presented on a computer)

SUMMARY:
This study aims to examine the effects of cognitive fatigue on heart rate variability and skin conductance and develop a machine learning model.

DETAILED DESCRIPTION:
We hypothesize that increased cognitive fatigue would vary as a function of heart rate variability and skin conductance. A machine learning model will be developed that predicts cognitive fatigue through these physiological responses (Lee et al., 2021). Individual differences (i.e., age, gender, caffeine and food intake, body mass index, skin temperature, sleep quality, baseline physiology and behavioural performance) will be examined and accounted for.

ELIGIBILITY:
Inclusion Criteria:

* Singapore-based
* Non-clinical
* 18-35years

Exclusion Criteria:

* Individuals with hearing difficulties or failing to meet the minimal threshold for normal hearing
* Individuals with a history of ear, developmental, neurological, or psychiatric disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 162 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
2-Back Task (Change) | during fatigue manipulation
  Change in Accuracy over time
2-Back Task (Change) | during fatigue manipulation
  Change in Reaction Time over time
Fatigue State Questionnaire | up to 5 mins after fatigue manipulation
  Fatigue State Questionnaire Score
Electrocardiograph (Change) | during fatigue manipulation
  Change in Heart Rate Variability over time
Electrodermal Activity (Change) | during fatigue manipulation
  Change in Skin Conductance Level over time
Electrodermal Activity (Change) | during fatigue manipulation
  Change in Skin Conductance Response over time

CONTACTS AND LOCATIONS:
Locations (1):
- Cultural Science Innovations, Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee KFA, Gan WS, Christopoulos G. Biomarker-Informed Machine Learning Model of Cognitive Fatigue from a Heart Rate Response Perspective. Sensors (Basel). 2021 Jun 2;21(11):3843. doi: 10.3390/s21113843. PMID 34199416